CLINICAL TRIAL: NCT00546533
Title: Open-Label Evaluation Of The Efficacy And Safety Of Etanercept In Patients With Active Rheumatoid Arthritis (RA)
Brief Title: Study Evaluating the Efficacy and Safety of Etanercept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A-101101
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
To assess the efficacy of etanercept 25 mg administered subcutaneously twice-weekly for 12 weeks in patients with active RA for whom classical antirheumatic therapy is insufficient or inappropriate.

ELIGIBILITY:
Inclusion Criteria:

* A negative serum or urine pregnancy test at screening and a medically acceptable form of contraception starting at screening and continuing throughout the study is required for all females of childbearing potential (defined as an oral, injectable, or implantable contraceptive, intrauterine device, or barrier method combined with a spermicide).
* Failed therapy with at least one DMARD (DMARD failure is defined as a discontinuation because of lack of clinical efficacy).
* Meet the 1987 American Rheumatism Association (ARA) revised criteria for rheumatoid arthritis.

Exclusion Criteria:

* Uncooperative patients with a history of poor compliance.
* Known hypersensitivity to etanercept or any of its components.
* Known significant concurrent medical disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-01; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To assess the clinical efficacy of etanercept 25 mg administered twice-weekly for 12 weeks in patients with active RA for whom classical antirheumatic therapy is insufficient or inappropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer